CLINICAL TRIAL: NCT02542631
Title: Glycemic Control and Treatment Satisfaction Using Finesse Versus Pen for Initiating Bolus Insulin Dosing in Type 2 Diabetes Mellitus Patients Not Achieving Glycemic Targets on Basal Insulin With/Without Anti-Hyperglycemic Agents
Brief Title: Glycemic Control and Treatment Satisfaction Using Finesse Versus Pen for Initiating Bolus Insulin Dosing in Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Calibra Medical, Inc. (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VP-00525; 2015-003761-28 (EudraCT Number)
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bolus Insulin Patch (Calibra Finesse) (Experimental): Use of the wearable patch to deliver meal-related bolus insulin dose
  Interventions: Device: Bolus Insulin Patch (Calibra Finesse)
- Insulin Pen (Novo-Nordisk FlexPen®) (Active Comparator): Use of the pen device to deliver meal-related bolus insulin dose
  Interventions: Device: Insulin Pen (Novo-Nordisk FlexPen®)

INTERVENTIONS:
Device: Bolus Insulin Patch (Calibra Finesse)
  Arms: Bolus Insulin Patch (Calibra Finesse)
Device: Insulin Pen (Novo-Nordisk FlexPen®)
  Arms: Insulin Pen (Novo-Nordisk FlexPen®)

SUMMARY:
To compare glycemic control and treatment satisfaction using a novel bolus insulin patch (Finesse) versus a pen for initiating and managing bolus insulin dosing in patients with T2DM not achieving glycemic targets on basal insulin with/without anti-hyperglycemic agents.

DETAILED DESCRIPTION:
Patients sub-optimally controlled on basal insulin (with/without other antihyperglycemic agents (AHAs)) will be randomized 1:1 to either Finesse or pen to initiate bolus insulin dosing and followed for a 44-week intervention period. Patients will have both basal and bolus doses of insulin adjusted throughout the trial, as is clinically indicated, based on an easy to follow insulin dosing algorithm. After the final endpoint evaluation at week 44, patients will crossover to the alternate bolus insulin delivery device for 4 weeks and complete a patient preference survey at week 48.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of T2DM
* Treated with basal insulin for ≥ 6 months, with current dose stable for ≥ 6 weeks of ≥ 0.3 U/kg/day, with or without anti-hyperglycemic agents and in whom the Investigator feels advancement from basal to basal and bolus therapy is needed for the patient
* A1C 7.5-11.0% by central lab value at screening visit
* Already perform self-monitoring of blood glucose (SMBG) and willing to test blood glucose (BG) over the course of the study
* Body Mass Index of ≤ 40 kg/m2

Exclusion Criteria:

* Currently on or has been treated in the past year with insulin regimens that include bolus insulins except the need for insulins in the settings of acute illness or hospitalization
* History of type 1 diabetes mellitus (T1DM), or diabetic ketoacidosis (DKA), or secondary forms of diabetes such as cystic fibrosis
* Known hypersensitivity or allergy to insulin-glargine or its excipients or any other insulins
* Two or more severe hypoglycemic episodes within the prior year
* Hypoglycemia unawareness defined by history
* History of proliferative diabetic retinopathy
* Is currently unstable and/or has moderate-to-severe medical illness in the Investigator's judgment
* Uncontrolled hypertension (either treated or untreated) defined as a systolic blood pressure ≥ 160 mmHg or a diastolic blood pressure ≥ 100 mmHg at screening
* History of recent major surgery within 6 months, or minor surgery within 3 months (such as appendectomy) prior to screening visit, or a planned surgery during the study period
* History of bariatric surgery
* Active chronic infections
* Women of child-bearing age who are pregnant, planning pregnancy, breast-feeding, or, if capable of pregnancy, are not practicing contraception if heterosexually active
* Known hypersensitivity to plastics/polymers/adhesives
* Known difficulties with adherence of adhesives, bandages, or dressings
* Participated in any research study within the past 30 days
* Currently participating in another investigational trial
* Use of short term or chronic systemic steroids within three months of entry into the study or likelihood that same might be required during the conduct of the study

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Bergenstal, MD, Principal Investigator — International Diabetes Center at Park Nicollet
Locations (52):
- United States (35):
  - Central Phoenix Medical Clinic, Phoenix, Arizona
  - Advanced Metabolic Care & Research Institute, Inc. (AMCR), Escondido, California
  - Marin Endocrine Care and Research, Greenbrae, California
  - National Research Institute - Wilshire, Los Angeles, California
  - Diabetes Research Institute Mills-Peninsula Health Service, San Mateo, California
  - Encompass Clinical Research, Spring Valley, California
  - Denver VA Medical Center, Denver, Colorado
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Physicians Research Associates, Lawrenceville, Georgia
  - Endocrine Research Solutions, Inc, Roswell, Georgia
  - Rocky Mountain Diabetes and Osteoporosis Center PA, Idaho Falls, Idaho
  - Northwestern University The Feinberg School of Medicine, Chicago, Illinois
  - John H. Stroger, Jr. Hospital of Cook County Diabetes Center, Chicago, Illinois
  - Iowa Diabetes and Endocrinology Research Center, Des Moines, Iowa
  - Cotton-O'Neil Clinical Research Center, Topeka, Kansas
  - Great Plains Diabetes, Wichita, Kansas
  - Kentucky Diabetes Endocrinology Center, Lexington, Kentucky
  - Medstar Health Research Institute, Hyattsville, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Park Nicollet Institute International Diabetes Center, Minneapolis, Minnesota
  - SUNY Upstate Medical University, Syracuse, New York
  - VA Medical Center Cleveland, Cleveland, Ohio
  - University Diabetes and Endocrine Consultants, Chattanooga, Tennessee
  - Texas Diabetes & Endocrinology, P.A.- Austin, Austin, Texas
  - Dallas Diabetes and Endocrine Center, Dallas, Texas
  - Baylor Endocrine Center, Dallas, Texas
  - Diabetes & Glandular Disease Clinic, P.A., San Antonio, Texas
  - South Texas Veterans Health Care System, San Antonio, Texas
  - Consano Clinical Research, San Antonio, Texas
  - Progressive Clinical Research, Bountiful, Utah
  - Highland Clinical Research, Salt Lake City, Utah
  - Danville Internal Medicine, Danville, Virginia
  - Private Practice-Larry Stonesifer, Federal Way, Washington
  - Rainier Clinical Research Center, Renton, Washington
- France (7):
  - Hopital Avicenne, Bobigny
  - Hopital Saint-Andre, Bordeaux
  - Hopital Hotel-Dieu Site Harfleur, Le Creusot
  - Lapeyronie Hospital, University Hospital Montpellier, Montpellier
  - Hopital Lariboisiere, Centre Universitaire du Diabete et de ses Complications, Paris
  - CHU de Nantes-Hospital Nord Laennec, Saint-Herblain
  - GHMP les Portes du Sud, Vénissieux
- Germany (3):
  - Diabeteszentrum DO-Diabetologisch, Dortmund
  - BAG Unterm Heilig Kreuz Unterm Heilig Kreuz, Fulda
  - Diabetes Zentrum und Praxis Prof. Pfutzner Parcusstr., Mainz
- United Kingdom (7):
  - Royal United Hospital, Diabetes & Lipid Research Wolfson Centre, Bath
  - Royal Blackburn Hospital, East Lancashire Hospitals NHS Trust, Blackburn
  - Chorley and South Ribble Hospital, Chorley
  - Ninewells Hospital & Medical School Diabetes Support Unit, Dundee
  - Forth Valley Royal Hospital Dept. of Diabetes, Larbert
  - Leicester General Hospital Leicester Diabetes Centre, Leicester
  - Royal Liverpool University Hospital, Liverpool

RESULTS

PARTICIPANT FLOW:
Groups:
- Bolus Insulin Patch: Experimental Treatment Arm
- Insulin Pen: Comparator Treatment Arm
Period: Overall Study
Arm/Group | Bolus Insulin Patch | Insulin Pen
Started (278) | 139 | 139
Completed (216) | 108 | 108
Not Completed | 31 | 31
Not completed — Adverse Event | 1 | 1
Not completed — Sponsor Termination | 1 | 0
Not completed — Withdrawal by Subject | 11 | 16
Not completed — Protocol Violation | 1 | 1
Not completed — Physician Decision | 6 | 4
Not completed — Lost to Follow-up | 6 | 5
Not completed — Death | 1 | 2
Not completed — Other | 2 | 1
Not completed — Used Prohibited Medication | 2 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Bolus Insulin Patch | Insulin Pen | Total
Number analyzed (Participants) | 139 | 139 | 278
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (9.7) | 60.4 (7.9) | 59.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 52 | 110
  Male | 81 | 87 | 168
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 4 | 1 | 5
  Black or African American | 12 | 11 | 23
  White | 120 | 126 | 246
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
A1C [Mean (Standard Deviation); unit: A1C %] — Baseline A1C Population: Intent-to-treat (ITT) population
  A1C % | 8.6 (0.9) | 8.7 (1.0) | 8.7 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in A1C From Baseline to the Completion of 24 Weeks of Basal and Bolus Insulin Therapy
Description: Change in A1C, with bolus insulin dosing with patch versus pen, from baseline to the completion of 24 weeks of basal and bolus insulin therapy
Time Frame: 24 weeks
Population: The primary outcome measure analysis used a modified intent-to-treat (mITT) population data set which included all the intent-to-treat (ITT) patients who had a baseline A1C and at least one post-baseline A1C measurement. For missing values, the last observation carried forward (LOCF) imputation method was used.
Measure: Least Squares Mean (Standard Error); unit: A1C %
Arm/Group | Bolus Insulin Patch | Insulin Pen
Number analyzed (Participants) | 136 | 138
A1C % | -1.69 (0.08) | -1.60 (0.08)
Statistical Analysis 1: Comparison: Bolus Insulin Patch vs Insulin Pen; Test type: Non-Inferiority — The sample size determination was based on the primary endpoint, A1C change from Baseline to Week 24. Assuming that the true mean difference in A1C change for Finesse versus Pen was -0.1% with a SD of 1.2%, a study population of 250 completers (125 per arm) was required to achieve a power of 90% for non-inferiority with a margin of 0.4%; p < 0.0001, ANCOVA — Non-inferiority p-value was calculated with 2-sided comparison of the difference in treatment effects between Finesse and Pen with a non-inferiority margin of 0.4%; ANCOVA model with treatment group as a factor and baseline value as a covariate was used to compare devices for continuous measures; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.32 to 0.14], Standard Error of Mean 0.12

2. Secondary Outcome: Number of Patients With A1C ≤7.0% at Week 24
Description: Number of patients with A1C ≤7.0% at week 24
Time Frame: 24 weeks
Population: Modified intent-to-treat (mITT) population data set.
Measure: Count of Participants; unit: Participants
Arm/Group | Bolus Insulin Patch | Insulin Pen
Number analyzed (Participants) | 136 | 138
Participants | 85 | 77
Statistical Analysis 1: Comparison: Bolus Insulin Patch vs Insulin Pen; Test type: Superiority; p = 0.26, Cochran-Mantel-Haenszel — Statistical test of device effects was conducted at a 2-sided alpha level of 0.05, and confidence interval (CI) was calculated at 95%, 2-sided; Odds Ratio (OR) = 1.3, 95% CI 2-sided [0.81 to 2.14], Standard Error of Mean 0.25

3. Secondary Outcome: Change in Percent of Glucose Values of Continuous Glucose Monitoring (CGM) Measurements Within Targeted Range of 71 and 180 mg/dl (4.0 and 10.0 mmol/l) From Baseline to Week 24
Description: Change in percent of glucose values of Continuous Glucose Monitoring (CGM) measurements within targeted range of 71 and 180 mg/dl (4.0 and 10.0 mmol/l) from baseline to week 24 (in a subset of patients)
Time Frame: 24 weeks
Population: Modified intent-to-treat population data subset.
Measure: Least Squares Mean (Standard Error); unit: % of glucose values
Arm/Group | Bolus Insulin Patch | Insulin Pen
Number analyzed (Participants) | 52 | 49
% of glucose values | 26.87 (2.33) | 29.84 (2.40)
Statistical Analysis 1: Comparison: Bolus Insulin Patch vs Insulin Pen; Test type: Superiority; p = 0.38, ANCOVA — [p-value comment as in outcome 2, analysis 1]; ACNOVA model with treatment group as a factor and baseline value as a covariate was used to compare devices for continuous measures; Mean Difference (Final Values) = -2.97, 95% CI 2-sided [-9.63 to 3.70], Standard Error of Mean 3.36

4. Secondary Outcome: Change in A1C From Baseline to Week 44
Description: Change in A1C from baseline to the completion of 44 weeks of basal and bolus insulin therapy
Time Frame: 44 weeks
Population: Only patients with non-missing baseline and endpoint values were included.
Measure: Least Squares Mean (Standard Error); unit: A1C %
Arm/Group | Bolus Insulin Patch | Insulin Pen
Number analyzed (Participants) | 108 | 109
A1C % | -1.63 (0.10) | -1.63 (0.10)
Statistical Analysis 1: Comparison: Bolus Insulin Patch vs Insulin Pen; Test type: Superiority; p = 0.99, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.28 to 0.28], Standard Error of Mean 0.14

5. Secondary Outcome: Number of Patients With A1C ≤7.0% at Week 44
Description: Number of patients with A1C ≤7.0% after 44 weeks of basal and bolus insulin therapy
Time Frame: 44 weeks
Population: Only patients with non-missing baseline and endpoint values were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Bolus Insulin Patch | Insulin Pen
Number analyzed (Participants) | 108 | 109
Participants | 70 | 68
Statistical Analysis 1: Comparison: Bolus Insulin Patch vs Insulin Pen; Test type: Superiority; p = 0.71, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.64 to 1.93], Standard Error of Mean 0.28

6. Secondary Outcome: Change in A1C From Week 24 to Week 44
Description: Change in A1C from week 24 to week 44 after basal and bolus insulin therapy
Time Frame: 44 weeks
Population: Only patients with non-missing week 24 and week 44 values were included.
Measure: Least Squares Mean (Standard Error); unit: A1C %
Arm/Group | Bolus Insulin Patch | Insulin Pen
Number analyzed (Participants) | 108 | 109
A1C % | 0.12 (0.06) | 0.07 (0.06)
Statistical Analysis 1: Comparison: Bolus Insulin Patch vs Insulin Pen; Test type: Superiority; p = 0.52, ANCOVA — [p-value comment as in outcome 2, analysis 1]; ANCOVA model with treatment group as a factor and week 24 value as a covariate was used to compare devices for continuous measures; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.12 to 0.24], Standard Error of Mean 0.09

7. Other Pre Specified Outcome: Change in Treatment Satisfaction From Baseline to Week 24
Description: Change in treatment satisfaction with insulin delivery system from baseline to week 24 was assessed by self-report on the validated Insulin Delivery System Rating Questionnaire. Scale is 0-100. Higher score is better.
Time Frame: 24 weeks
Population: Per Protocol. Only patients with non-missing baseline and endpoint values were included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Bolus Insulin Patch | Insulin Pen
Number analyzed (Participants) | 124 | 117
units on a scale | 13.63 (1.94) | 4.47 (2.01)
Statistical Analysis 1: Comparison: Bolus Insulin Patch vs Insulin Pen; Test type: Superiority; p = 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; ANCOVA model with change in score as dependent variable, treatment as factor, and baseline score as a covariate was used to compare devices; Mean Difference (Final Values) = 9.16, 95% CI 2-sided [3.65 to 14.67], Standard Error of Mean 2.80

8. Other Pre Specified Outcome: Change in Quality of Life From Baseline to Week 24
Description: Change in Diabetes-Specific Quality of Life (QOL), baseline to week 24. was assessed by self-report on the validated Diabetes Specific Quality of Life Survey. Scale is 0-100. Higher score is better.
Time Frame: 24 weeks
Population: Per Protocol. Only patients with non-missing baseline and endpoint values were included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Bolus Insulin Patch | Insulin Pen
Number analyzed (Participants) | 124 | 123
units on a scale | 2.37 (1.43) | -1.95 (1.44)
Statistical Analysis 1: Comparison: Bolus Insulin Patch vs Insulin Pen; Test type: Superiority; p = 0.03, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 4.32, 95% CI 2-sided [0.33 to 8.32], Standard Error of Mean 2.03

9. Secondary Outcome: Number of Participants With Severe Hypoglycemic Event
Description: An event requiring the assistance of another person to actively administer carbohydrate (including IV dextrose), glucagon, or other resuscitative actions. Neurological recovery attributable to the restoration of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration.
Time Frame: 44 weeks
Population: Intent to Treat. All patients randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Bolus Insulin Patch | Insulin Pen
Number analyzed (Participants) | 139 | 139
Participants | 3 | 3
Statistical Analysis 1: Comparison: Bolus Insulin Patch vs Insulin Pen; Test type: Superiority; p = 1.00, Chi-squared

ADVERSE EVENTS:
Time Frame: 44 weeks
Description: A SAE is an event that led to death, or serious deterioration in health that either resulted in a life-threatening illness or injury, or permanent impairment of a body structure or body function, or in-patient hospitalization or prolongation of existing hospitalization, or medical or surgical intervention to prevent life threatening illness or injury or permanent impairment to a body structure or body function; or that led to fetal distress, fetal death or congenital abnormality or birth defect.
Arm/Group | Bolus Insulin Patch | Insulin Pen
All-Cause Mortality (participants affected / at risk) | 1/139 | 2/139
Serious Adverse Events (participants affected / at risk) | 10/139 | 13/139
Other Adverse Events (participants affected / at risk) | 100/139 | 99/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bolus Insulin Patch (N=139) | Insulin Pen (N=139)
Cardiac disorders (Cardiac disorders) | 5 (7) | 2 (2)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 (2) | 2 (3)
General Disorders (General disorders) | 2 (3) | 0 (0)
Infections and Infestations (Infections and infestations) | 0 (0) | 3 (3)
Nervous system disorders (Nervous system disorders) | 1 (1) | 2 (2)
Vascular disorders (Vascular disorders) | 1 (1) | 2 (2)
Neoplasms benign, malignant, and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1) | 0 (0)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bolus Insulin Patch (N=139) | Insulin Pen (N=139)
General disorders (General disorders) | 28 (39) | 15 (15)
Respiratory, thoracic, and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 14 (18) | 17 (22)
Nervous system disorders (Nervous system disorders) | 13 (15) | 16 (19)
Investigations (Investigations) | 10 (10) | 14 (14)
Vascular disorders (Vascular disorders) | 12 (12) | 8 (9)
Infections and infestations (Infections and infestations) | 51 (84) | 60 (85)
Musculoskeletal and connective tissue (Musculoskeletal and connective tissue disorders) | 34 (48) | 32 (42)
Gastrointestinal disorders (Gastrointestinal disorders) | 23 (37) | 21 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT02542631/Prot_SAP_000.pdf